CLINICAL TRIAL: NCT02020902
Title: Contac Bien Z Adverse Effect Survey
Brief Title: Post Marketing Surveillance for Contac Bien Z in Japan
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 200638; RH01905 (Other: GSK)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Allergic Rhinitis; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cetrizine hydrochloride — As provided on the patient information leaflet

SUMMARY:
This is a post-marketing surveillance study on a marketed cetrizine hydrochloride formulation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, between 15-65 years of age, who purchase the marketed cetrizine hydrochloride formulation

Exclusion Criteria:

* Who have ever experienced allergic symptoms by taking this medication or any component of this medication, piperazine derivative (including levocetirizine, hydroxizine)
* Those who have been under 15en diagnosed with kidney disease
* Children under 15 years of age

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who purchase the marketed cetrizine hydrochloride formulation from pharmacy stores in Japan.
Sampling Method: Probability Sample
Enrollment: 1552 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adverse events after having cetrizine hydrochloride | At baseline
  Participants will answer a questionnaire which consists of questions on safety of the marketed cetrizine hydrochloride formulation.

SECONDARY OUTCOMES:
Efficacy of the marketed cetrizine hydrochloride formulation | At baseline
  Participants will answer a questionnaire which consists of questions on their satisfaction after taking the marketed cetrizine hydrochloride formulation. The efficacy will be measured on a 4 point scale (1 Efficacious; 2 Somewhat efficacious; 3 Not efficacious; 4 Not known)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Drug Store Seki, Saitama, Japan